CLINICAL TRIAL: NCT04744870
Title: Tissue Monitoring During Endovascular Intervention
Acronym: TIME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pedra Technology, PTE LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-002
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease; Arterial Occlusive Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Tissue perfusion assessment is key to more accurate measurement of foot ischemia, which is in turn an important factor in appropriate treatment decisions. In practice though, tissue perfusion measurements are not routinely undertaken as few practical solutions exist that are easy to use and fit in everyday clinical practice. Pedra has developed a novel, easy to use, non-invasive device that can be used in practice to better inform treatment decisions.

DETAILED DESCRIPTION:
Tissue perfusion assessment is key to more accurate measurement of foot ischemia, which is in turn an important factor in appropriate treatment decisions. In practice though, tissue perfusion measurements are not routinely undertaken as few practical solutions exist that are easy to use and fit in everyday clinical practice. Pedra has developed a novel, easy to use, non-invasive device that can be used in practice to better inform treatment decisions.

This is a feasibility study to demonstrate the ability of the Xauron system to track tissue perfusion changes in patients undergoing endovascular intervention for the treatment of peripheral artery disease (PAD). The findings of this study are for research purposes and will also be used to help with the future education of physicians about the potential use of the Xauron system. In addition, this early pilot data will be used to help power larger, more definitive studies relating to the intra-procedural use of the Xauron system.

ELIGIBILITY:
Inclusion Criteria:

* The subject is undergoing endovascular intervention for the management of their PAD.
* The subject is between 40 and 90 years of age.
* Documented lower limb arterial occlusive or stenotic disease (using ankle-brachial index / pulse volume recording, duplex ultrasound or CT angiogram) within the last 8 weeks.
* In the opinion of the Investigator, the subject is willing and able to comply with the protocol and complete all protocol assessments.
* Subject has been informed of the nature of the study, agrees to its provisions and has willingly provided written informed consent, approved by the appropriate Institutional Review Board (IRB)

Exclusion Criteria:

* Subjects on an investigational drug or being treated with an investigational therapeutic device, within 30 days of the study visit, that in the view of the Investigator might interfere with the study outcomes.
* Presence of a condition that the Investigator considers will compromise the subject's ability to participate in the study.
* Subjects on renal replacement therapy
* Signs of active infection causing localized inflammation on the plantar or dorsal surfaces of the foot.
* Diabetic subjects with a Charcot neuropathic osteoarthropathy
* Lack of intact skin, or pathological skin conditions, at the proposed sensor pad positions that may impair or prevent the adherence of medical adhesives in general.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, multi-center, observational, feasibility study to collect tissue perfusion data throughout the duration of a standard of care (SOC) endovascular intervention, alongside live video capture of the angiography utilized during the case. The study will enroll up to 80 subjects between the ages of 40 and 90 who are undergoing endovascular intervention for the management of their PAD. The protocol is designed for sites to enroll approximately half of the subjects with primary "below the knee disease".
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Integration of Xauron System into clinical workflow - The Investigator will complete a questionnaire assessing that the Xauron system can be integrated within the angiography suite for all subjects observed. | Measured at the SOC index procedure
  To confirm that the Xauron system can be integrated into the angiography suite clinical workflow.

SECONDARY OUTCOMES:
Relationship between interventional events of procedure and perfusion changes detected by Xauron System | Measured at the SOC index procedure
  Measure the time from end of an intervention to the zenith or nadir of the subsequent perfusion change
Relationship of perfusion data from different anatomical locations during procedure | Measured at the SOC index procedure
  Determine the ratio of perfusion in the arm relative to the foot after an intervention
User feedback from the team in the angiographic suite | Measured at the SOC index procedure
  To obtain user feedback from the team in the angiography suite, to improve the user interface between the device and the operators.
Relationship between changes in perfusion during intervention and the clinical outcomes of patients using the Walking Score. | Measured through 3-month follow-up
  Evaluate the relationship between changes in perfusion during the intervention and the clinical outcomes of the patients in terms of changes in the Walking Score.
Angiographic images to evaluate and understand perfusion monitoring | Measured at the SOC index procedure
  Collate data and angiographic images/video that may help endovascular teams understand and utilize perfusion monitoring in the angiography suite.
Relationship between changes in perfusion during intervention and the clinical outcomes of patients using the Pain Score. | Measured through 3-month follow-up
  Evaluate the relationship between changes in perfusion during the intervention and the clinical outcomes of the patients in terms of changes in the Pain Score.
Relationship between changes in perfusion during intervention and the clinical outcomes of patients using the SF-36 Score | Measured through 3-month follow-up
  Evaluate the relationship between changes in perfusion during the intervention and the clinical outcomes of the patients in terms of changes in the SF-36 score.